CLINICAL TRIAL: NCT01810757
Title: A Multicentre Randomised Phase II Study of HYpofractionated Bladder Radiotherapy With or Without Image Guided aDaptive Planning
Brief Title: Study of Weekly Radiotherapy for Bladder Cancer
Acronym: HYBRID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR3973; CRUK/12/055 (Other Grant/Funding Number: CRUK); ICR-CTSU/2013/10039 (Other: ICR-CTSU Protocol Number)
Record Dates: First submitted 2013-03-08; First posted 2013-03-14 (Estimated); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard planning (Active Comparator): Standard planning radiotherapy
  Interventions: Radiation: Standard planning radiotherapy
- Adaptive planning (Experimental): Adaptive planning radiotherapy
  Interventions: Radiation: Adaptive planning radiotherapy

INTERVENTIONS:
Radiation: Standard planning radiotherapy — 36 Gray dose given in 6 fractions of 6 Grays over 6 weeks, using one plan per patient.
  Arms: Standard planning
Radiation: Adaptive planning radiotherapy — 36 Gray dose given in 6 fractions of 6 Grays over 6 weeks, selecting the best fit from three plans per patient.
  Arms: Adaptive planning

SUMMARY:
Background Localised muscle invasive bladder cancer (MIBC) is life-threatening and can cause significant symptoms. Around 50% of patients with MIBC who are referred for radiotherapy are unfit for standard radical treatment (surgery or daily radiotherapy with chemotherapy), but would have a normal life expectancy if their cancer were adequately controlled. Retrospective studies suggest that radiotherapy which is given weekly using fewer fractions and higher doses (hypofractionated), may be an alternative where daily radiotherapy is not an option.

Radiotherapy treatment is planned based on information from a CT scan which shows the position and shape of the bladder. This plan needs to take into account the fact that the bladder's shape and position can change, depending on how full it is and because of where it is in relation to the bowel. A safety margin is therefore added around the bladder on the planned treatment, to reduce the risk of missing any of the bladder with the radiotherapy.

It is now possible to take scans of the bladder's position before each treatment and adjust the position of the treatment plan accordingly to ensure the bladder is fully covered by it. In this study we are also looking at whether it is possible to design a series of treatment plans with different size safety margins and then choose one that fits best for each particular day. This is called 'adaptive radiotherapy'. This technique may enable accurate treatment delivery using smaller safety margins and this might help to reduce side effects.

Aims

In patients with MIBC not suitable for cystectomy or daily radiotherapy we aim to assess:

1. whether treatment using adaptive planning can be successfully delivered at multiple sites across the UK and results in acceptable levels of toxicity
2. the local tumour control rate achieved by hypofractionated weekly radiotherapy
3. the requirement to treat with adaptive planning.

How results will be used Results will provide robust evidence for use of hypofractionated radiotherapy and assess whether this is a plausible and worthwhile treatment in this patient population. The randomised element of the trial will support the implementation of image-guided adaptive radiotherapy for bladder cancer in the UK. HYBRID will provide evidence on the benefits or otherwise of this methodology and inform the development of further trials in this and other patient groups.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary To assess whether adaptive radiotherapy techniques when delivered at multiple centres can lead to a reduction in the level of acute non-genitourinary (GU) toxicity experienced by patients with muscle invasive bladder cancer unsuitable for daily radical radiotherapy.

Secondary

* Establish the local disease control rates of hypofractionated bladder radiotherapy as measured at 3 months
* Assess time to local disease progression
* Assess the overall survival time of patients who have received hypofractionated radiotherapy.
* Investigate the control rate of presenting symptoms, the effect of hypofractionated treatment on late radiotherapy side effects and patient reported outcomes.
* To establish the proportion of fractions benefiting from adaptive planning.

OUTLINE: This is a multicentre randomised Phase II study in patients with muscle invasive bladder who are not suitable for cystectomy or daily radiotherapy.

All patients will be planned to receive six 6Gray (Gy) fractions of image guided radiotherapy delivered weekly (total dose: 36Gy) and will be randomised to standard or adaptive planning.

Participants allocated to the standard planning group will have one radiotherapy plan generated and this will be used to deliver all 6 treatments, with a cone beam CT scan prior to treatment delivery which can be used by the local investigator to adjust treatment delivery according to local practice.

Participants allocated to adaptive planning will have three radiotherapy plans generated; small, medium and large. A cone beam CT taken prior to each treatment delivery will be used to select the most appropriate plan of the day.

Patients are followed up in terms of the trial up to 24 months, after this time only basic routine follow-up data will be collected.

PROJECTED ACCURAL: The aim is to recruit 62 participants, 31 to each treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Histologically confirmed invasive bladder carcinoma (T2-T4a N0 M0; any histological sub-type)
* Unsuitable for radical cystectomy or daily fractionated radiotherapy for any reason (including performance status, co-morbidity, patient refusal)
* Expected survival >6 months
* WHO performance status 0-3
* Willing to undergo post treatment cystoscopy

Exclusion Criteria:

* Nodal or metastatic disease
* Concurrent malignancy
* Previous pelvic radiotherapy
* Urinary catheter in-situ
* Any other contra-indication to radiotherapy (e.g. inflammatory bowel disease)
* Unable to attend for post treatment follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2023-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Huddart, Principal Investigator — Institute of Cancer Research/RMNHSFT
Locations (11):
- United Kingdom (11):
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Ipswich Hospital, Ipswich
  - St James's University Hospital, Leeds
  - Guy's & St Thomas's Hospital, London
  - Royal Marsden NHSFT, London
  - University College London, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich
  - Royal Preston Hospital, Preston
  - Queens Hospital, Romford

REFERENCES:
- [Result] Farbiszewski R, Ustymowicz J, Dudek H. [Participation of free radicals in the mechanism of brain tissue damage]. Neurol Neurochir Pol. 1993 Sep-Oct;27(5):729-37. Polish. PMID 8114997
- [Derived] Hafeez S, Patel E, Webster A, Warren-Oseni K, Hansen V, McNair H, Miles E, Lewis R, Hall E, Huddart R. Protocol for hypofractionated adaptive radiotherapy to the bladder within a multicentre phase II randomised trial: radiotherapy planning and delivery guidance. BMJ Open. 2020 May 26;10(5):e037134. doi: 10.1136/bmjopen-2020-037134. PMID 32461298

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Planning | Adaptive Planning
Started | 32 | 33
Completed | 32 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Planning | Adaptive Planning | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 84.8 [80.7 to 88.9] | 84.1 [80.4 to 87.1] | 84.5 [80.6 to 88.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 24 | 20 | 44
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 33 | 65
Extent of resection [Count of Participants; unit: Participants]
  Biopsy | 10 | 10 | 20
  Partial resection | 10 | 13 | 23
  Full resection | 11 | 9 | 20
  Unobtainable | 1 | 1 | 2
Multiple tumours [Count of Participants; unit: Participants]
  Yes | 6 | 7 | 13
  No | 26 | 26 | 52
Histological tumour type [Count of Participants; unit: Participants]
  Urothelial | 31 | 32 | 63
  Non-urothelial | 1 | 1 | 2
Grade [Count of Participants; unit: Participants] — higher grade is worse as tissue is less normal like
  Participants
    Grade 1 | 0 | 0 | 0
    Grade 2 | 1 | 0 | 1
    Grade 3 | 31 | 33 | 64
Carcinoma in situ (CIS) present [Count of Participants; unit: Participants]
  Yes | 9 | 11 | 20
  No | 22 | 22 | 44
  Unobtainable | 1 | 0 | 1
Clinical stage [Count of Participants; unit: Participants] — Describes the size of the tumour. A higher clinical T stage is worse.
  Participants
    T1 | 0 | 0 | 0
    T2 | 24 | 21 | 45
    T3a | 1 | 5 | 6
    T3b | 5 | 5 | 10
    T4a | 2 | 2 | 4
Age adjusted Charlson Comorbidity index score [Count of Participants; unit: Participants] — Age-adjusted Charlson comorbidity index is used to predict the risk of mortality in patients with multiple comorbidities. A higher score is worse and the score ranges from 0-37
  Participants
    5 | 1 | 0 | 1
    6 | 14 | 13 | 27
    7 | 11 | 5 | 16
    8 | 4 | 6 | 10
    9 | 2 | 8 | 10
    10 | 0 | 0 | 0
    11 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Experiencing Severe Acute Non-genitourinary Side Effects Following Radiotherapy.
Description: Non-GU CTCAE G3+ treatment-related toxicity occurring within the first 3 months of radiotherapy completing
Time Frame: 12 weeks from completion of radiotherapy
Population: Evaluable patient population: This population contains all randomised patients who have received at least one fraction of radiotherapy and are evaluable for the primary endpoint of acute toxicity (i.e. toxicity reported up to 3 months post radiotherapy). Patients had been reviewed for evaluability by the independent Trial steering committee (TSC) blinded to planning method and the TSC's view on evaluability for the primary endpoint has been used to define the evaluable patient population.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Planning | Adaptive Planning
Number analyzed (Participants) | 30 | 33
Participants | 4 | 2

2. Secondary Outcome: Local Disease Control Rate
Description: Presence of cancer in the bladder 3 months after treatment. Presented as the proportion of all patients regardless of treatment allocation (standard and adaptive combined) having evidence of residual tumour.
Time Frame: 3 months
Population: Including only those who had an assessment at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Planning | Adaptive Planning
Number analyzed (Participants) | 23 | 25
Participants | 17 | 22

3. Secondary Outcome: Time to Local Disease Progression
Description: From randomisation to a maximum follow-up of 30 months. It was pre-planned in the SAP to combine the two treatment arms together because there is insufficient statistical power to detect clinically meaningful differences.
Time Frame: Event-free survival estimates at 12 months and 24 months are reported.
Population: Intention to treat population. It was pre-planned in the SAP to combine the two treatment arms together because there is insufficient statistical power to detect clinically meaningful differences.
Measure: Number (95% Confidence Interval); unit: percentage event-free
Groups:
- Overall: Including the standard and adaptive arms
Arm/Group | Overall
Number analyzed (Participants) | 65
percentage event-free
  KM 12 months | 71.7 [55.9 to 82.6]
  KM 24 months | 47.3 [29.6 to 63.1]

4. Secondary Outcome: Overall Survival
Description: From randomisation to maximum follow-up of 56 months. It was pre-planned in the SAP to combine the two treatment arms together because there is insufficient statistical power to detect clinically meaningful differences.
Time Frame: Event-free survival estimates at 12 months and 24months are reported.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage surviving
Groups:
- Overall: Includes standard and adaptive patients
Arm/Group | Overall
Number analyzed (Participants) | 65
percentage surviving
  KM 12 months | 61.5 [48.6 to 72.1]
  KM 24 months | 46.2 [33.8 to 57.7]

5. Secondary Outcome: The Control Rate of Presenting Symptoms
Description: Assessed by looking at change in symptom scores from pre to post radiotherapy. The number of patients with post-radiotherapy scores lower than their baseline score have been used to calculate the control rate of presenting symptoms and is presented separately for the two randomisation groups.
Time Frame: 3 months from the completion of radiotherapy
Population: Including those with 3 month follow up acute toxicity available. Frequency threshold for reporting: Renal and urinary symptom reported in 20% or more of patients with symptoms/toxicity reported.
Measure: Number; unit: participants
Arm/Group | Standard Planning | Adaptive Planning
Number analyzed (Participants) | 27 | 29
participants
  Cystitis | 3 | 8
  Haematuria | 4 | 8
  Nocturia | 3 | 5
  Frequency/Urgency | 5 | 7
  Urinary incontinence | 4 | 4

6. Secondary Outcome: The Proportion of Fractions Benefiting From Adaptive Planning
Description: Assessed by the number of small or large plans being selected rather than the medium plan for patients in the adaptive planning group. The denominator will be the total number of fractions received in the adaptive planning group.
Time Frame: End of treatment, treatment is given over 6 weeks
Population: ITT
Measure: Count of Units; unit: Fractions
Units Other Than Participants: Fractions
Arm/Group | Adaptive Planning
Number analyzed (Participants) | 33
Number analyzed (Fractions) | 193
Fractions | 76

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 24 months.
Description: Adverse event data were collected at the following timepoints:
  Baseline Acute toxicity: RT week1, RT week2, RT week3, RT week4, RT week5, RT week6, Post RT week4, Post RT 3M Late toxicity: 6M, 12M, 24M
Arm/Group | Standard Planning | Adaptive Planning
Serious Adverse Events (participants affected / at risk) | 11/32 | 9/33
Other Adverse Events (participants affected / at risk) | 32/32 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Planning (N=32) | Adaptive Planning (N=33)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 4 (4)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Planning (N=32) | Adaptive Planning (N=33)
Abdominal pain (Gastrointestinal disorders) | 13 (35) | 15 (42)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 8 (27) | 6 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (11) | 1 (2)
Bladder obstruction (Renal and urinary disorders) | 11 (34) | 7 (8)
Bladder pain (Renal and urinary disorders) | 1 (3) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 15 (41) | 9 (17)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin decreased (Investigations) | 1 (3) | 0 (0)
Blood creatinine increased (Investigations) | 14 (62) | 10 (28)
Blood phosphorus decreased (Investigations) | 1 (5) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 2 (4)
Blood sodium decreased (Investigations) | 1 (2) | 0 (0)
Blood urea increased (Investigations) | 3 (11) | 3 (13)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chills (General disorders and administration site conditions) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 22 (96) | 16 (58)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cystitis (Renal and urinary disorders) | 21 (63) | 21 (77)
Decreased appetite (Metabolism and nutrition disorders) | 17 (57) | 16 (51)
Dehydration (Metabolism and nutrition disorders) | 6 (9) | 9 (34)
Diarrhoea (Gastrointestinal disorders) | 23 (50) | 22 (64)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (8) | 4 (17)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders and administration site conditions) | 31 (188) | 31 (168)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (4) | 2 (8)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 17 (44) | 16 (46)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hot flush (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (6) | 4 (7)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (6) | 3 (5)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 3 (4)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (14) | 8 (24)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 28 (193) | 31 (209)
Non-cardiac chest pain (General disorders and administration site conditions) | 1 (1) | 0 (0)
Pelvic pain (Renal and urinary disorders) | 2 (2) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 28 (175) | 30 (182)
Proctitis (Gastrointestinal disorders) | 6 (9) | 5 (7)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (2) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (7) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (2) | 3 (12)
Urinary incontinence (Renal and urinary disorders) | 16 (62) | 19 (75)
Urinary retention (Renal and urinary disorders) | 3 (11) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (8) | 6 (12)
Urinary tract obstruction (Renal and urinary disorders) | 2 (4) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 7 (11)
Weight decreased (Investigations) | 10 (24) | 9 (14)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes